CLINICAL TRIAL: NCT00592592
Title: A Phase II Trial of Proton RT for the Treatment of Pediatric Rhabdomyosarcoma
Brief Title: Proton Radiation Therapy (RT) for the Treatment of Pediatric Rhabdomyosarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Brigham and Women's Hospital (Other); Boston Children's Hospital (Other); Dana-Farber Cancer Institute (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Torunn Yock, MD, Director, Pediatric Radiation Oncology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-188; P01CA021239 (NIH)
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Rhabdomyosarcoma
Keywords: pediatric rhabdomyosarcoma; proton radiation therapy
MeSH Terms: conditions — Rhabdomyosarcoma | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Beam Radiation (Experimental): Proton Beam Radiation
  Interventions: Radiation: Proton Beam Radiation

INTERVENTIONS:
Radiation: Proton Beam Radiation — Once per day, 5 days a week for a total of 4 to 6 weeks.

SUMMARY:
The main purpose of this study is to see if using proton beam radiation therapy instead of photon beam radiation therapy can reduce side effects from radiation treatment for rhabdomyosarcoma. Photon beam radiation is the standard type of radiation for treating most rhabdomyosarcoma and many other types of cancer. Photon beam radiation enters the body and passes through healthy tissue, encounters the tumor, then leaves the body through healthy tissue. A beam of proton radiation enters the body and passes through healthy tissue, encounters tumor, but then stops. This means that less healthy tissue is affected by proton beam radiation than by photon beam radiation.

DETAILED DESCRIPTION:
* A special device is made for each participant to help them hold still during the treatment. This may be in the form of a mask or a custom made foam cradle depending on the area to be treated.
* Radiation treatments will be given once per day, 5 days a week for a total of 4 to 6 weeks, depending upon how much total dose the tumor requires.
* Participants will be seen once per week by their radiation doctor to monitor health and record any side effects from treatment.
* After the radiation treatments are completed, participants will be required to undergo further tests and evaluations for several years following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven newly diagnosed rhabdomyosarcoma.
* Patients less than or equal to 30 years of age.
* Patients must be treated with a standardly accepted chemotherapy regimen.
* May not have metastatic disease unless aged 2-10 with embryonal histology.
* Must be willing to receive follow-up care for a minimum of five years after treatment at MGH and annual visits unless it is too difficult to return to MGH for follow-up care. In that event, they must be willing to have their outside medical information released to us to track the results.
* Timing of radiation must be according to the IRB protocol upon which the patient is treated within either 35 days of last chemotherapy or surgery.

Exclusion Criteria:

* Life expectancy of less than 2 years.
* Co-morbidities that would make the use of radiation too toxic to deliver safely, such as serious local injury or collagen vascular disease.
* Patients who are pregnant
* Previous treatment with radiation therapy.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torunn Yock, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Preliminary results of a phase II trial of proton radiotherapy for pediatric rhabdomyosarcoma — http://www.ncbi.nlm.nih.gov/pubmed/25332253

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Beam Radiation
Started | 115
Completed | 114
Not Completed | 1
Not completed — Patient found ineligible upon chart review | 1

BASELINE CHARACTERISTICS:
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 114
Age, Continuous [Mean (Full Range); unit: years] — Patient aged 24.6 was granted an exception by the IRB and included in the study despite being over 21.
  years | 4.3 [0.6 to 24.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 86
  More than one race | 0
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  United States | 114

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence (Estimated Percent of Participants) With Grade 3 or Higher Toxicity in Follow-up
Description: Cumulative incidence of participants who experienced a toxicity defined as either grade 3, 4, or 5 after the completion of radiation therapy in pediatric patients with pediatric rhabdomyosarcomas. Late toxicity is scored on a yearly follow-up basis for at least five years. Late toxicities will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0. Cumulative incidence is shown at 5 years follow-up.
Time Frame: 5 years from the start of radiation treatment
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 114
Percentage of patients | 10.9 [5.7 to 18.0]
Statistical Analysis 1: Comparison: Proton Beam Radiation; Test type: Other; Cumulative incidence = 10.9, 95% CI 2-sided [5.7 to 18.0]

2. Secondary Outcome: Percentage of Participants Who Experienced an Acute Toxicity by Grade
Description: Percentage of participants who experienced an acute toxicity following completion of radiation treatment by grade. Acute toxicity will be scored at weekly status check visits by the radiation oncology nurse or doctor. In addition, acute toxicity will be scored at least one time within the 3 months following completion of radiation therapy. The recommended evaluation time for acute toxicity after radiotherapy was 6 weeks following completion, but may be at any time during the 3 months after treatment. Acute toxicities are graded according to the Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0. Toxicities are graded on a scale of 1 to 5. A higher grade indicates a worse outcome with 1 being mild, 4 being life-threatening, and 5 being death.
Time Frame: 3 months from radiation treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 114
Participants
  Grade 1 | 110
  Grade 2 | 92
  Grade 3 | 30
  Grade 4 | 5
  Grade 5 | 0

3. Secondary Outcome: Dosimetric Comparison
Description: Comparison of dose distribution to tumor and surrounding normal structures using dose volume histograms (DVH) generated from the proton plan used to treat the patient and the photon plan generated for comparison purposes. Percent of normal tissue spared was calculated using the following equation: (100 x (mean x-ray dose - mean proton dose))/mean X-ray dose. No measure of dispersion was calculated for these estimates. The data is no longer available.
Time Frame: 4 years from the start of radiation treatment
Population: Patients who had DVH's generated from proton plans for comparison
Measure: Number; unit: Percentage of normal tissue spared of RT
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 54
Percentage of normal tissue spared of RT
  Hypothalamus | 88
  Pituitary | 73
  Lens (Contra) | 100
  Maxilla | 42
Statistical Analysis 1: Comparison: Proton Beam Radiation; Test type: Other; p < 0.01, t-test, 2 sided; Paired t-test; % hypothalamus normal tissue spared = 88
Statistical Analysis 2: Comparison: Proton Beam Radiation; Test type: Other; p < 0.01, t-test, 2 sided; Paired t-test; % pituitary normal tissue spared = 73
Statistical Analysis 3: Comparison: Proton Beam Radiation; Test type: Other; p < 0.01, t-test, 2 sided; Paired t-test; % lens (contra) normal tissue spared = 100
Statistical Analysis 4: Comparison: Proton Beam Radiation; Test type: Other; p = 0.02, t-test, 2 sided; Paired t-test; % maxilla normal tissue spared = 42

4. Secondary Outcome: Local Control
Description: Estimated survival probability (defined as being free of a local recurrence) was calculated using Grays formula for competing risks
Time Frame: 5 years from the start of radiation therapy
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 114
percent probability | 80.9 [73.0 to 87.7]
Statistical Analysis 1: Comparison: Proton Beam Radiation; Test type: Other; Percent Survival, Local Control = 80.9, 95% CI 2-sided [73.0 to 87.7]

ADVERSE EVENTS:
Time Frame: All adverse events, both serious and non-serious, and deaths were collected from the initiation of study intervention, during treatment, and annually for at least 5 years from the start of radiation treatment.
Description: Acute toxicity was scored at weekly status check visits by the radiation oncology nurse or doctor. In addition, acute toxicity was scored at least one time within the 3 months following completion of radiation therapy. Late toxicity were scored on a yearly follow-up basis for at least five years. Adverse events were monitored through study completion. Toxicities are graded according to the Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0.
Arm/Group | Proton Beam Radiation
All-Cause Mortality (participants affected / at risk) | 28/114
Serious Adverse Events (participants affected / at risk) | 6/114
Other Adverse Events (participants affected / at risk) | 113/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton Beam Radiation (N=114)
Right eye blindness (Eye disorders) | 1 — Grade 4, Unrelated to study treatment
Abdominal pain (Gastrointestinal disorders) | 1 — Grade 3, Unrelated to study treatment
Mood alteration- Depression (Psychiatric disorders) | 1 — Grade 4, Unrelated to study treatment
Infection- Other (Thrush) (Infections and infestations) | 1 — Grade 2, Definitely related to study treatment
Infection- Other (C Diff) (Infections and infestations) | 1 — Grade 3. Unrelated to study treatment.
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 — Grade 4, Unrelated to study treatment
Dehydration (Metabolism and nutrition disorders) | 1 — Grade 3. Probably related to study treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton Beam Radiation (N=114)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 9
Hearing w/w-o audiogr in monitor prg (Ear and labyrinth disorders) | 11
Hearing-other (Ear and labyrinth disorders) | 9
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 7
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 3
Hearing w/o audiogr not in monitor prg (Ear and labyrinth disorders) | 1
Hemoglobin (Investigations) | 8
Neutrophils (Investigations) | 8
Leukocytes (Investigations) | 6
Lymphopenia (Blood and lymphatic system disorders) | 4
Hematologic-other (Blood and lymphatic system disorders) | 4
Platelets (Investigations) | 3
Fatigue (General disorders) | 66
Weight loss (Metabolism and nutrition disorders) | 9
Constitutional, other (General disorders) | 2
Fever w/o neutropenia (General disorders) | 1
Odor (patient odor) (General disorders) | 1
Radiation dermatitis (Injury, poisoning and procedural complications) | 89
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 42
Erythema multiforme (Skin and subcutaneous tissue disorders) | 21
Skin-other (Skin and subcutaneous tissue disorders) | 20
Alopecia (Skin and subcutaneous tissue disorders) | 5
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Atrophy, Subcutaneous fat (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Induration/fibrosis (Skin and subcutaneous tissue disorders) | 2
Athropy, skin (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 1
Injection site reaction (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1
Growth hormone secretion abnormality (Endocrine disorders) | 11
Hypothyroidism (Endocrine disorders) | 9
Endocrine-other (Endocrine disorders) | 5
Adrenal insufficiency (Endocrine disorders) | 3
Gonadotropin secretion abnormality (Endocrine disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 40
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 40
Nausea (Gastrointestinal disorders) | 26
Vomiting (Gastrointestinal disorders) | 17
Taste disturbance (Gastrointestinal disorders) | 13
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 12
Teeth (Gastrointestinal disorders) | 11
Teeth development (Gastrointestinal disorders) | 11
Dysphagia (Gastrointestinal disorders) | 10
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 9
GI-other (Gastrointestinal disorders) | 7
Dehydration (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 3
Muco/stomatitis by exam, pharynx (Gastrointestinal disorders) | 3
Salivary (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Fistula, Oral Cavity (Gastrointestinal disorders) | 1
Incontinence, anal (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, rectum (Gastrointestinal disorders) | 1
Ulcer, anus (Gastrointestinal disorders) | 1
Growth velocity reduction (Endocrine disorders) | 9
Short stature (Musculoskeletal and connective tissue disorders) | 4
Limb length discrepancy (Musculoskeletal and connective tissue disorders) | 3
Puberty, precocious (Endocrine disorders) | 2
Alteration in bone age (Musculoskeletal and connective tissue disorders) | 1
Spine kyphosis/lordosis (Musculoskeletal and connective tissue disorders) | 1
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 11
Hemorrhage-other (General disorders) | 3
Anus, hemorrhage (Gastrointestinal disorders) | 1
Rectum, hemorrhage (Gastrointestinal disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Infection-other (Infections and infestations) | 32
Infection w/ unk ANC conjunctiva (Infections and infestations) | 2
Infection w/ unk ANC oral cavity/gums (Infections and infestations) | 2
Infection w/ unk ANC sinus (Infections and infestations) | 2
Infection Gr0-2 neut, conjunctiva (Infections and infestations) | 1
Infection Gr0-2 neut, sinus (Infections and infestations) | 1
Edema head and neck (Blood and lymphatic system disorders) | 17
Lymphatics-other (Blood and lymphatic system disorders) | 1
Edema limb (Blood and lymphatic system disorders) | 1
Muscular/skeletal hypoplasia (Musculoskeletal and connective tissue disorders) | 36
Trismus (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 7
Joint-function (Musculoskeletal and connective tissue disorders) | 3
Bone: spine-scoliosis (Musculoskeletal and connective tissue disorders) | 2
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 2
Nonneuropathic facial muscle weak (Musculoskeletal and connective tissue disorders) | 2
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 2
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 13
Anxiety (Psychiatric disorders) | 11
Irritability (children < 3yrs of age) (Psychiatric disorders) | 4
Dizziness (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 2
Neuropathy CN III pupil/eyelid/extraocul (Nervous system disorders) | 2
Neurologic-other (Nervous system disorders) | 2
Neuropathy CN VII face-motor / taste (Nervous system disorders) | 1
Neuropathy CN IX pharynx ear tongue (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 1
Speech impairment (Nervous system disorders) | 1
Ocular-other (Eye disorders) | 38
Cataract (Eye disorders) | 22
Dry eye syndrome (Eye disorders) | 16
Tearing (Eye disorders) | 10
Vision-blurred (Eye disorders) | 9
Ocular surface disease (Eye disorders) | 6
Eyelid dysfunction (Eye disorders) | 5
Proptosis/enophthalmos (Eye disorders) | 5
Keratitis (Eye disorders) | 4
Vision-photophobia (Eye disorders) | 4
Nystagmus (Eye disorders) | 2
Double vision (Eye disorders) | 2
Retinopathy (Eye disorders) | 1
Scleral necrosis/melt (Eye disorders) | 1
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 21
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 5
Urinary frequency/urgency (Renal and urinary disorders) | 5
Incontinence urinary (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 3
Renal/GU-other (Renal and urinary disorders) | 2
Cystitis (Renal and urinary disorders) | 1
Sexual/Reproductive function-Other (Reproductive system and breast disorders) | 2
Vascular-Other (Specify) (Vascular disorders) | 2
Vessel injury Carotid (Vascular disorders) | 1
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 15
Oral cavity, pain (Gastrointestinal disorders) | 14
Pain-other (General disorders) | 9
Eye, pain (Eye disorders) | 7
Head/headache (Nervous system disorders) | 7
Face, pain (General disorders) | 5
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 3
Middle ear, pain (Ear and labyrinth disorders) | 3
Abdomen, pain (Gastrointestinal disorders) | 2
Back, pain (Musculoskeletal and connective tissue disorders) | 2
Neck, pain (Musculoskeletal and connective tissue disorders) | 2
Oral gums, pain (Gastrointestinal disorders) | 2
Rectum, pain (Gastrointestinal disorders) | 2
Anus, pain (Gastrointestinal disorders) | 1
Buttock, pain (Musculoskeletal and connective tissue disorders) | 1
Esophagus, pain (Gastrointestinal disorders) | 1
External ear, pain (Ear and labyrinth disorders) | 1
Liver, pain (Hepatobiliary disorders) | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1
Ovulatory, pain (Reproductive system and breast disorders) | 1
Pelvic, pain (Reproductive system and breast disorders) | 1
Pain NOS (General disorders) | 1
Urethra, pain (Renal and urinary disorders) | 1
Vagina, pain (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes